CLINICAL TRIAL: NCT07019064
Title: A Phase 1, Randomized, Open-label, Single-dose, Crossover, Relative Bioavailability Study of Omaveloxolone Intact Capsules Versus Capsule Contents Sprinkled Over Low-fat, Non-Greek Yogurt in Healthy Adult Subjects
Brief Title: A Study to Learn How BIIB141 (Omaveloxolone) is Processed in the Body When Taken as Capsules Compared to Sprinkled on Yogurt in Healthy Adults Aged 18 to 55
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 296HV103
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — omaveloxolone

STUDY DESIGN:
Intervention Model Description: This 2-way crossover study will be conducted in 2 Periods with a washout period of 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive treatment A (omaveloxolone capsule orally on Day 1) followed by treatment B (omaveloxolone capsule content sprinkled over low-fat, non-Greek yogurt on Day 15).
  Interventions: Drug: Omaveloxolone
- Treatment Sequence BA (Experimental): Participants will receive treatment B (omaveloxolone capsule content sprinkled over low-fat, non-Greek yogurt on Day 1) followed by treatment A (omaveloxolone capsule orally on Day 15).
  Interventions: Drug: Omaveloxolone

INTERVENTIONS:
Drug: Omaveloxolone — Administered as specified in the treatment arm.
  Other Names: BIIB141

SUMMARY:
In this study, researchers will learn more about how BIIB141, also known as omaveloxolone or SKYCLARYS®, is processed in the body when taken in different ways. This drug has been approved, or made available for doctors to prescribe, for people with Friedrich's Ataxia (FA) who are at least 16 years old. Currently, people with FA can take it either as whole capsules or opening the capsules and sprinkling its contents over applesauce. The main goal of this study is to learn if BIIB141 is processed any differently when taken sprinkled over low-fat, non-Greek yogurt compared to whole capsules. This will help researchers learn if yogurt could be another option for people to take BIIB141 with.

The main questions researchers want to answer in this study are :

• How does the body process BIIB141 when taken as whole capsules compared to being sprinkled over yogurt?

Researchers will also learn more about :

* How many participants have adverse reactions during the study. An adverse reaction is a health problem that may be caused by the study drug.
* If there are any changes in the participants' overall health during the study

This study will be done as follows:

* Participants will be screened to check if they can join the study. The screening period will be up to 28 days, after which participants will check into their study research center.
* Participants will stay at the study research center for about 30 days.
* This is a "crossover" study. In this kind of study, all participants receive the same 2 or more study drugs (or ways of taking the drug), but the order in which they receive them depends on the group they are randomly assigned to.
* In Group 1, participants will take a single dose of BIIB141 as a capsule, followed by a break of 14 days. Then, the participants will take a single dose of BIIB141 sprinkled over yogurt.
* In Group 2, participants will take a single dose of BIIB141 sprinkled over yogurt, followed by a break of 14 days. Then, the participants will take a single dose of BIIB141 as a capsule.
* Each participant will be in the study for up to 57 days.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the relative bioavailability of omaveloxolone capsules when administered as either intact capsules or capsule contents sprinkled over low-fat, non-Greek yogurt in healthy adult participants. The secondary objective of the study is to evaluate the safety and tolerability of a single dose of omaveloxolone administered as either an intact capsule or sprinkled over low-fat, non-Greek yogurt in healthy adult participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Body Mass Index (BMI) at screening between 18 and 32 kilograms per meter square (kg/m^2), inclusive
* Must be in good health as determined by the Investigator, based on medical history and Screening evaluations

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease
* History of, or ongoing, malignant disease (with exceptions for completely excised basal cell carcinomas and squamous cell carcinomas cured at least 1 year prior to Day -1)
* Systolic blood pressure > 150 millimeters of mercury (mmHg) or < 90 mmHg after sitting for 5 minutes
* Clinically significant, as determined by the Investigator, 12-lead electrocardiogram (ECG) abnormalities
* Corrected QT interval > 450 milliseconds (ms) for males and > 460 ms for females
* Positive diagnostic tuberculosis test result within 30 days of Enrollment
* History of, or positive test result for human immunodeficiency virus (HIV)
* History of hepatitis C infection or positive test result for hepatitis C virus antibody (HCV Ab)
* Current hepatitis B infection
* Any value for alanine aminotransferase, aspartate aminotransferase, bilirubin, or serum creatinine above the upper limit of normal
* Platelets below the lower limit of normal
* Any clinically significant value out of normal range for total white blood cells
* Prior exposure to the study treatment
* Use of prescription medication (excluding oral contraceptives and hormone replacement therapy), over-the-counter oral medication that alters hepatic or renal clearance, or nutraceuticals within 28 days prior to Day -1
* Use of other over-the-counter oral medication, vitamins, dietary supplements, or antacids within 14 days prior to Day -1

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Omaveloxolone | Pre-dose and at multiple time points post dose up to Day 29
Area Under the Concentration-Time Curve From Time Zero to Time of the Last Measurable Concentration (AUC0-t) of Omaveloxolone | Pre-dose and at multiple time points post dose up to Day 29
Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Omaveloxolone | Pre-dose and at multiple time points post dose up to Day 29

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to end of study (up to 29 days)
Number of Participants with Abnormalities in Clinical Laboratory Assessments, Vital Signs, and Electrocardiogram (ECGs) | From Day 1 up to end of study (up to 29 days)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Trialmed formerly PPD, Austin Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/